CLINICAL TRIAL: NCT05811754
Title: Post-marketing Commitment Safety Study of HZ/su to Evaluate Pregnancy Exposures and Outcomes in Immunodeficient or Immunosuppressed Women Between 18 and 49 Years of Age
Brief Title: Safety of Herpes Zoster Subunit (HZ/su) Vaccine During Pregnancy in Adult Women With Immunocompromised Conditions
Status: Active, not recruiting | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Harvard Pilgrim Health Care Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 214420
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-08

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Recombinant; Zoster vaccine; Targeted; Safety study; Post-authorization safety study; Pregnant women
MeSH Terms: conditions — Herpes Zoster | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HZ/su-Exposed Group: Pregnancies among adult women diagnosed with immunocompromised conditions who were exposed to the HZ/su vaccine during pregnancy.
  Interventions: Other: Data collection
- Comparison (Unexposed) Group: Pregnancies among adult women diagnosed with immunocompromised conditions who were not exposed to the HZ/su vaccine during pregnancy.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — This study will be conducted using data provided by U.S. Research Partners in the FDA's Sentinel Surveillance System.
  Four Research Partners will participate in this study: CVS Health Clinical Trial Services (CTS), Carelon Research, Optum and Harvard Pilgrim Health Care Institute (HPHCI).

SUMMARY:
The purpose of this post-marketing commitment safety study is to evaluate the real-world safety of HZ/su vaccine during pregnancy in immunodeficient or immunosuppressed adult pregnant women between 18 and 49 years of age in the United States. The primary outcome of interest is major congenital malformations (MCMs).

ELIGIBILITY:
Inclusion Criteria:

* Participant who is pregnant with a pregnancy start date between 01 July 2021 and 30 June 2026. Live births are to be followed for 1 year.
* Participant is a female aged 18-49 years on the pregnancy start date.
* Participant meets study definition of systemic lupus erythematosus (SLE), multiple sclerosis (MS), rheumatoid arthritis (RA), inflammatory bowel disease (IBD), psoriasis (PsO)/psoriatic arthritis (PsA), solid organ transplant (SOT), stem cell transplant (SCT), hematologic malignancies (HM), solid tumors (ST), or human immunodeficiency virus (HIV). Codes for immunocompromised conditions will be identified in the health plan claims of the Distributed Research Network (DRN) during the period 273 days prior to the pregnancy start date through the first trimester (98 days after the pregnancy start date). Diagnoses recorded through the first trimester will be included to account for women who may not have frequent visits prior to pregnancy and may have a more complete assessment of medical conditions during the first prenatal care visit.
* Participant has at least 273 days of continuous health plan enrollment with medical and drug benefits prior to the start of pregnancy through the delivery date, with gaps of up to 45 days in coverage being permitted. The 273-day pre-pregnancy period through the first trimester (a period of 98 days after the pregnancy start date) was chosen to allow identification of potential confounders of interest. In Sentinel projects, gaps of 45 days or less in health plan enrolment are typically considered administrative gaps (and not lapses in health plan coverage) and ignored.

Exclusion Criteria:

* Participant was exposed to a medication(s) that presents a known increased risk for fetal malformations.
* Participant delivered an infant identified as having a chromosomal or genetic anomaly.
* Ectopic pregnancies, molar pregnancies or induced abortions.
* Multigestation (e.g., twin) pregnancies.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Adult pregnant women, 18-49 years of age, diagnosed with an immunocompromised condition who were members of any of the 4 participating Sentinel Research Partners.
Sampling Method: Probability Sample
Enrollment: 2844 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Major Congenital Malformations (MCMs) | From birth up to 1 year of age
  The prevalence of MCMs among live births from women with immunocompromised conditions exposed to HZ/su vaccine compared to those not exposed to HZ/su vaccine during pregnancy is evaluated.
  An MCM (birth defect or structural defect) is defined as a defect, which has either cosmetic or functional significance to the child.

SECONDARY OUTCOMES:
Prevalence of additional infant/birth outcomes (small for gestational age, low birthweight, neonatal intensive care unit admission) | Within 30 days after the infant's date of birth
  The prevalence of small for gestational age, low birthweight, neonatal intensive care unit admission among live births in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.
Prevalence of additional infant/birth outcome (preterm birth) | At birth
  The prevalence of the preterm births among live births in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.
Prevalence of additional infant/birth outcome (neonatal death) | Within 28 days after birth
  The prevalence of the neonatal deaths among live births in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.
Prevalence of pregnancy outcomes (live birth) | At birth
  The prevalence of the live birth pregnancies among all eligible pregnancies in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.
Prevalence of pregnancy outcomes (stillbirth) | At or after 20 weeks' gestation but prior to delivery
  The prevalence of the stillbirth pregnancies among all eligible pregnancies in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.
Prevalence of pregnancy outcomes (spontaneous abortion) | Prior to 20 weeks' gestation
  The prevalence of the spontaneous abortions among all eligible pregnancies in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.
Prevalence of pregnancy complications | From 20 weeks' gestation through the date of delivery
  The prevalence of pregnancy complications (placental abruption, preeclampsia and eclampsia) among livebirth and non-livebirth pregnancies in women with immunocompromised conditions exposed to HZ/su vaccine versus those not exposed to HZ/su vaccine during pregnancy is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Canton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No